CLINICAL TRIAL: NCT06994884
Title: Patients' Experiences of Information After Total Knee Arthroplasty - A Qualitative Interview Study
Status: Not yet recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: 283839
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Knee Osteoarthrosis; Total Knee Arthroplasty
Keywords: total knee arthroplasty; qualitative research; knee osteoarthrosis; primary care; physical therapy specialty
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Interview group: To ensure variation in the sample, diversity in age and sociodemographic background is sought.
  Inclusion criteria: Men and women of all ages who have undergone total knee arthroplasty due to osteoarthritis and are undergoing rehabilitation in primary care.
  Exclusion criteria: Previous joint replacement in the hip or knee.

SUMMARY:
The aim of this qualitative interview study is to gain new and in-depth knowledge about patients' experiences of information following total knee arthroplasty. Participants will be interviewed in the recovery phase after surgery. Researchers will use a semi-structured interview guide. The interviews will be analysed with qualitative content analysis.

DETAILED DESCRIPTION:
A qualitative interview study will be conducted. Interviews will be conducted 24-28 weeks after total knee arthroplasty. A semi-structured interview guide will be used to answer the following research questions:

* What are the patients' positive and negative experiences of the information provided before and after total knee arthroplasty (TKA)?
* What are the patients' experiences and perceptions regarding the content and scope of the information, as well as how and when it is communicated?
* What are the patients' experiences and perceptions of their access to information?
* What are the patients' experiences and perceptions of the significance of the information for postoperative care and their expectations of the surgical outcome?
* How do patients perceive the information provided before and after surgery in relation to their expectations of the information?
* How do patients think the information provided before and after TKA could be improved?

ELIGIBILITY:
Inclusion Criteria:

* Men and women of all ages who have undergone total knee arthroplasty due to osteoarthritis and are undergoing rehabilitation in primary care.

Exclusion Criteria:

* Previous joint replacement in the hip or knee.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from two hospitals in Region Västra Götaland, Sweden. Mölndal Hospital is located in the city of Gothenburg, while Alingsås Hospital is situated in the smaller city of Alingsås and also serves a rural population.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-08-18 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Qualitative content analysis | Interviews will be performed 24-28 weeks after total knee arthroplasty
  The transcribed interviews will be analyzed in their entirety using qualitative content analysis, which includes interpretation of the manifest content of the text as well as a deeper interpretation of the underlying latent meaning. First, the transcripts will be read repeatedly to gain a sense of the whole. Then, meaning units that respond to the study's aim will be identified from the text, without being separated from their context. In the next step, these units will be condensed to shorten the text while preserving its core content. Based on the condensed meaning units, subcategories, categories, and themes will be formed by moving back and forth between the whole text and its parts. Potential subcategories, categories, and themes will be discussed within the research team until consensus is reached, in order to enhance the credibility of the analysis. The results will be presented as themes, categories, and/or subcategories.

IPD SHARING:
Plan to Share IPD: Undecided